CLINICAL TRIAL: NCT02319603
Title: A Randomized, Double-blind, Two Dose Group, Parallel-control Multi-center, Post-marketing Clinical Trial,to Evaluate the Efficacy and Safety of Wenxin Keli in Treating Atrial Premature Beats.
Brief Title: To Evaluate the Efficacy and Safety of Wenxin Keli in Treating Atrial Premature Beats
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Bozhiyin T&S Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WX-20141022
Record Dates: First submitted 2014-12-02; First posted 2014-12-18 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Premature Beats
MeSH Terms: conditions — Atrial Premature Complexes | interventions — wenxin keli

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose WenXin keli (Active Comparator): Low dose group (the original quantity Wenxin keli): specification 10g /bag, Wenxin keli (no sugar) 5 g+ Wenxin keli simulation agent 5g.
  Oral ,1 bag each time, 3 times a day, 4 weeks for 1 course of treatment.
  Interventions: Drug: Low dose WenXin keli
- High dose WenXin keli (Experimental): High dose group(2 times the amount of Wenxin keli): specification 10g /bag, Wenxin keli (no sugar) 10 g.
  Oral ,1 bag each time, 3 times a day, 4 weeks for 1 course of treatment.
  Interventions: Drug: High dose WenXin keli

INTERVENTIONS:
Drug: Low dose WenXin keli — Low dose WenXin keli (the original quantity Wenxin keli): specification 10g /bag, Wenxin keli (no sugar) 5 g+ Wenxin keli simulation agent 5g.
  Other Names: the original quantity Wenxin keli
  Arms: Low dose WenXin keli
Drug: High dose WenXin keli — High dose WenXin keli(2 times the amount of Wenxin keli): specification 10g /bag, Wenxin keli (no sugar) 10 g.
  Other Names: 2 times the amount of Wenxin keli
  Arms: High dose WenXin keli

SUMMARY:
A randomized, double-blind, two dose group, parallel-control multi-center, post-marketing clinical trial，to evaluate the efficacy and safety of Wenxin keli in treating atrial premature beats by different dose,to provide a scientific basis for rational clinical use of drug.

DETAILED DESCRIPTION:
Research purpose： To evaluate the efficacy and safety of Wenxin keli in treating atrial premature beats by different dose,to provide a scientific basis for rational clinical use of drug.

Research design： A randomized, double-blind, two dose group, parallel-control multi-center, post-marketing clinical trial.

Sample size:

A total of 288 subjects, 144cases in each group.

Therapeutic schedule:

1. Low dose group (the original quantity Wenxin keli): specification 10g /bag, Wenxin keli (no sugar) 5 g+ Wenxin keli simulation agent 5g.
2. High dose group(2 times the amount of Wenxin keli): specification 10g /bag, Wenxin keli (no sugar) 10 g.

Usage and Dosage:

Oral ,1bag each time, 3 times a day, 4 weeks for 1 course of treatment.

Drug combination:

During the test shall not merge the other anti-arrhythmic drugs beyond the provisions of this scheme. Due to merger disease or condition changes ,have to use drugs or other treatment, investigators must record the types (or other treatment ),drug usage, time and reasons, in order to summarize ,analyze and report.

Primary indicator:

24 h dynamic electrocardiogram (Holter): before treatment, after treatment of 4 w, each record at a time.

Secondary Indicator:

Symptom scores: before treatment, after treatment of 4 w, each record at a time.

Security index:

1. Vital signs: before treatment, after treatment of 4 w, each record at a time.
2. Blood, urine, stool occult blood ,liver and kidney function, blood coagulation four, electrolyte examination, electrocardiogram(ecg): before treatment, after treatment of 4 w, each record at a time.

Main efficacy:

Holter efficient curative effect (main efficacy index) Effective: premature beat frequency reduced 50% or more before taking the medicine.

Invalid: no effective standard.

Secondary efficacy:

Symptom scores curative effect Effective:symptoms improve symptoms(drop 1or above) Invalid: no effective standard.

Statistic analysis:

Main efficacy index by means of FAS,PPS analysis ,safety index SS set analysis.

ELIGIBILITY:
Inclusion Criteria:

* Accord with the diagnostic criteria of arrhythmia (atrial premature beats )
* The average number of premature beat of 24 h dynamic electrocardiogram >360 times/h (effective record at least 22 h)
* Stop using the anti- arrhythmic drugs for more than five half-life (except that who long-term (one month or more) with beta blockers for high blood pressure and exertional angina)
* Ages 18 to 75 years old ,all genders
* Voluntary subjects and signed the informed consent form

Exclusion Criteria:

* Need to merge other anti-arrhythmic drugs(Ⅰ,Ⅱ,Ⅲ,Ⅳ) for serious condition
* Heart rhythm disorders caused by the factors such as drugs ,electrolyte and acid-base balance disorders
* Merge tardy arrhythmia (including sick sinus syndrome and Ⅱdegree atrioventricular block)
* Patients have had heart percutaneous coronary intervention (PCI) and coronary artery bypass grafting (CABG) surgery
* Patients with severe hypotension
* With serious cardiovascular diseases (severe coronary heart disease, congenital heart disease, cardiomyopathy, myocardial infarction, congestive heart failure, cardiac shock, etc.), cerebrovascular disease, severe respiratory diseases (chronic obstructive pulmonary disease, pulmonary hypertension, pulmonary embolism, etc.),serious primary diseases such as liver, kidney and hematopoietic system (ALT,AST,BUN 2 times higher than normal ceiling, or Cr higher than the upper limit of normal)
* Allergic constitution; the test drug allergy or its ingredients or elements allergy
* Pregnancy and lactation women ,recent preparation pregnancy
* With chronic alcoholism , drug dependence, mental illness
* Participated in other clinical trials within 3 months
* Patients thought by the investigators not suitable to participate in clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
24 h dynamic electrocardiogram (Holter) | Baseline, up to 4 weeks, each record at a time.
  Baseline, up to 4 weeks, each record at a time.

SECONDARY OUTCOMES:
Symptom scores | Baseline, up to 4 weeks, each record at a time.
  Baseline, up to 4 weeks, each record at a time.

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Guo, doctor, Principal Investigator — Director of department
Locations (1):
- Peking University people's hospital, Beijing, Beijing Municipality, China